CLINICAL TRIAL: NCT01979354
Title: The Comparison of 0.15 Milligram Spinal Morphine vs.no Treatment for Morphine Requirement After Video-assisted Thoracoscopic Surgery. A Pilot Randomized Control Study
Brief Title: 0.15 mg Spinal Morphine vs. no Treatment for Morphine Requirement After VATs.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sirilak Suksompong, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 552/2556(EC3)
Record Dates: First submitted 2013-11-02; First posted 2013-11-08 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Postoperative Pain
Keywords: spinal morphine; VATs lobectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spinal morphine (Active Comparator): 0.15 mg spinal morphine
  Interventions: Drug: Spinal morphine
- Control (No Intervention): No spinal morphine

INTERVENTIONS:
Drug: Spinal morphine — 0.15 mg spinal morphine
  Arms: Spinal morphine

SUMMARY:
Postoperative pain after Video-assisted Thoracoscopic Surgery (VAT) is still debating. Therefore the investigators conduct a study comparing 0.15 mg spinal morphine and control group in term of analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 year or over
* Patient ASA physical status I-III.
* Scheduled for video-assisted thoracoscopic lobectomy or blebectomy with pleurectomy or pleural abrasion
* Can operate a patient-controlled analgesia (PCA) device.

Exclusion Criteria:

* Known hypersensitivity to morphine
* History of bleeding tendency.
* Known case of infection at the back
* Patient refuse for spinal anesthesia
* History of cerebrovascular disease.
* Need mechanical ventilatory support during postoperative period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Total morphine requirement in 48 hours | 48 hours

SECONDARY OUTCOMES:
Pain | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Principal Investigator — Mahidol University
Locations (1):
- Mahidol University, Bangkok, Thailand